CLINICAL TRIAL: NCT02342678
Title: Lessening Incontinence Through Low-impact Activity, a.k.a. Yoga to Enhance Behavioral Self-Management of Urinary Incontinence in Women
Brief Title: Lessening Incontinence Through Low-impact Activity
Acronym: LILA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-14732; 1R34AT008028-01A1 (NIH)
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Yoga; Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yoga Therapy Group (Experimental): Participants will take part in twice weekly group yoga classes focusing on selected Iyengar-based yoga techniques as well as practice study-specific yoga techniques at home for at least one hour per week for a total of 12 weeks. During a 12-week post-treatment follow-up period, participants will also be encouraged to continue practicing yoga exercises for at least an hour per week.
  Interventions: Behavioral: Yoga Therapy
- Physical Conditioning Group (Experimental): Patricipants will take part in twice weekly group physical conditioning classes and practice stretching exercises at least one hour per week at home for 12 weeks. During a 12-week post-treatment follow-up period, participants will also be encouraged to continue practicing stretching exercises for at least an hour per week.
  Interventions: Behavioral: Physical Conditioning

INTERVENTIONS:
Behavioral: Yoga Therapy
  Arms: Yoga Therapy Group
Behavioral: Physical Conditioning
  Arms: Physical Conditioning Group

SUMMARY:
The LILA study is a pilot randomized parallel-group trial of a group-based yoga therapy program versus physical conditionin control program for treatment of urinary incontinence in ambulatory middle-aged and older women. Women aged 50 years and older who meet the criteria for frequency of incontinence episodes, are not using other clinical treatments for incontinence, and meet minimum physical mobility requirements and other eligibility criteria will be recruited from the general San Francisco Bay Area.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50 years or older who report urinary incontinence starting at least 3 months prior to screening
* Self-report at least required frequency of urinary incontinence episodes on a screening 3-day voiding diary
* Self-report urgency-predominant (i.e., at least half of incontinence episodes being urgency-type), stress-predominant (i.e., at least half of episodes being stress-type), or mixed-type (i.e., an equal number of stress- and urgency-type episodes) incontinence on the screening voiding diary
* Willing to refrain from initiating medical treatments that may affect their incontinence or voiding pattern during the study intervention period

Exclusion Criteria:

* Participation in formal or organized yoga classes or instruction within the past 3 months; or any prior yoga therapy directed specifically at improving urinary incontinence or pelvic floor dysfunction
* Participation in at least weekly organized physical conditioning classes or instruction in the past 3 months involving muscle stretching and strengthening exercises (not including aerobic classes that do not emphasize stretching or strengthening).
* Currently pregnant (by self-report or screening urine pregnancy test), gave birth within the past 6 months, or planning pregnancy during the study period (approximately 2 to 6 months)
* Current urinary tract infection (screening dipstick urinalysis with leukocyte estrace, nitrites or blood) or a history or 3 or more urinary tract infections in the preceding year
* Report history of neurologic conditions such as stroke, multiple sclerosis, spinal cord injury, or Parkinson's disease, or a lumbosacral spine condition associated with neurological symptoms
* Unable to walk up a flight of stairs or at least 2 blocks on level ground without assistance (i.e., functional capacity < 4 METs)
* Unable to get up from a supine to a standing position in 10 seconds or less and without assistance
* Morbid obesity defined by a measured body mass index of >40 kg/m2 at the screening evaluation.
* Report any history of prior anti-incontinence or urethral surgery (not including urethral dilation), pelvic cancer, or pelvic irradiation for any reason
* Report use of bladder botox, electrostimulation, bladder training, or pelvic floor exercise training (with certified practitioners) in the past 3 months
* Report other surgery to the pelvis (hysterectomy, oophorectomy, vaginal surgery, bladder surgery, colon surgery) within the past 3 months
* Report use of medications with the potential to affect incontinence (anticholinergic bladder medications, tricyclic antidepressants, selective norepinephrine reuptake inhibitors, mirabegron, loop diuretics) within the past month
* Report starting stopping, or changing the dose of a medication with the potential to affect anxiety or stress symptoms (i.e., selective serotonin reuptake inhibitors, anxiolytics/sedatives, antipsychotics) within the past 1 month, or plans to start, stop, or change to dose of such a medication during the study period
* Report use of medical devices (i.e. pessary) for incontinence within the previous month (participants may stop use of device and re-present for study)
* Report history of interstitial cystitis, fistula or hole in bladder or rectum, or birth defect leading to urine leakage
* Report symptomatic pelvic organ prolapse (assessed using a standardized question, ""Have your pelvic organs (uterus, bladder, or rectum) been dropping out of your vagina causing a feeling of bulging, pressure, or protrusion or a sensation like your "insides are coming out"?")
* Report history of vulvodynia, chronic pelvic pain, or pain when practicing pelvic floor exercises
* Report conditions that, in the judgment of the investigators, render potential participants unlikely to follow the protocol, including plans to move, substance abuse, significant psychiatric problems, or dementia
* Participation in another research study that involves investigational drugs or devices that could potentially confound the results of this study
* Unable to understand study procedures, complete study interviews, or and provide informed consent in English

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison J Huang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Nicosia FM, Lisha NE, Chesney MA, Subak LL, Plaut TM, Huang A. Strategies for evaluating self-efficacy and observed success in the practice of yoga postures for therapeutic indications: methods from a yoga intervention for urinary incontinence among middle-aged and older women. BMC Complement Med Ther. 2020 May 14;20(1):148. doi: 10.1186/s12906-020-02934-3. PMID 32408868
- [Derived] Huang AJ, Chesney M, Lisha N, Vittinghoff E, Schembri M, Pawlowsky S, Hsu A, Subak L. A group-based yoga program for urinary incontinence in ambulatory women: feasibility, tolerability, and change in incontinence frequency over 3 months in a single-center randomized trial. Am J Obstet Gynecol. 2019 Jan;220(1):87.e1-87.e13. doi: 10.1016/j.ajog.2018.10.031. Epub 2018 Oct 26. PMID 30595143

RESULTS

PARTICIPANT FLOW:
Groups:
- Yoga Therapy Group: Participants will take part in twice weekly group yoga classes focusing on selected Iyengar-based yoga techniques as well as practice study-specific yoga techniques at home for at least one hour per week for a total of 12 weeks. During a 12-week post-treatment follow-up period, participants will also be encouraged to continue practicing yoga exercises for at least an hour per week.
  Yoga Therapy
- Physical Conditioning Group: Patricipants will take part in twice weekly group physical conditioning classes and practice stretching exercises at least one hour per week at home for 12 weeks. During a 12-week post-treatment follow-up period, participants will also be encouraged to continue practicing stretching exercises for at least an hour per week.
  Physical Conditioning
Period: Overall Study
Arm/Group | Yoga Therapy Group | Physical Conditioning Group
Started | 28 | 28
Completed | 27 | 23
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Too busy to complete study | 0 | 2
Not completed — Family illness/emergency | 0 | 1
Not completed — Illness/medical reason | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga Therapy Group | Physical Conditioning Group | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 12 | 28
  >=65 years | 12 | 16 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Latina White | 18 | 17 | 35
  Latina White | 1 | 1 | 2
  Asian/Asian-American | 4 | 6 | 10
  Native Hawaiian or Pacific Islander | 2 | 2 | 4
  Unknown | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56
Incontinence Frequency [Mean (Standard Deviation); unit: Episodes per day]
  Total Incontinence | 3.8 (1.6) | 3.1 (2.3) | 3.5 (2.0)
  Urgency Incontinence | 2.1 (1.8) | 2.3 (2.3) | 2.2 (2.1)
  Stress Incontinence | 1.4 (1.5) | 0.7 (1.1) | 1.0 (1.4)
Urinary Symptom Questionnaire Scores [Mean (Standard Deviation); unit: Scores on Scale]
  Incontinence Impact Questionnaire | 117.9 (82.1) | 133.9 (92.3) | 125.9 (87.0)
  Urogenital Distress Inventory-6 | 34.5 (16.4) | 36.5 (19.5) | 35.5 (17.8)
  Patient Perception of Bladder Condition | 3.4 (1.0) | 3.3 (1.1) | 3.4 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Total Incontinence Frequency
Description: Change in the frequency of urinary incontinence episodes of any type. Analysis of covariance models were developed to examine change in incontinence frequency over 3 months. Results were summarized using least square mean estimates of changes in incontinence frequency in each group, as well as estimates of between-group difference in change in outcomes. Main efficacy analyses included all participants regardless of drop-out or adherence, consistent with an intention-to-treat principle. To address the potential for bias stemming from missing bladder diary data for up to 16% of participants who dropped out of interventions early, a multiple imputation procedure (SAS PROC MI, SAS Institute, Inc.) was used to impute values for data missing at follow-up. Imputation models included outcomes, randomization group, and baseline values.
Time Frame: Baseline and 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes per day
Arm/Group | Yoga Therapy Group | Physical Conditioning Group
Number analyzed (Participants) | 28 | 28
episodes per day | -2.8 [-3.6 to -2.0] | -1.9 [-2.8 to -0.9]
Statistical Analysis 1: Comparison: Yoga Therapy Group vs Physical Conditioning Group; Test type: Superiority; p = 0.13, ANCOVA; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-0.3 to 2.2]

2. Secondary Outcome: Stress-type Incontinence Frequency
Description: Change in the frequency of stress-type incontinence episodes Analysis of covariance models were developed to examine change in incontinence frequency over 3 months. Results were summarized using least square mean estimates of changes in incontinence frequency in each group, as well as estimates of between-group difference in change in outcomes. Main efficacy analyses included all participants regardless of drop-out or adherence, consistent with an intention-to-treat principle. To address the potential for bias stemming from missing bladder diary data for up to 16% of participants who dropped out of interventions early, a multiple imputation procedure (SAS PROC MI, SAS Institute, Inc.) was used to impute values for data missing at follow-up. Imputation models included outcomes, randomization group, and baseline values.
Time Frame: Baseline and 3 Months
Measure: Least Squares Mean (95% Confidence Interval); unit: Episodes per day
Arm/Group | Yoga Therapy Group | Physical Conditioning Group
Number analyzed (Participants) | 28 | 28
Episodes per day | -0.8 [-1.2 to -0.4] | -0.4 [-0.9 to 0.1]
Statistical Analysis 1: Comparison: Yoga Therapy Group vs Physical Conditioning Group; Test type: Superiority; p = 0.18, ANCOVA; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.2 to 1.1]

3. Secondary Outcome: Urgency-type Incontinence
Description: Change in frequency of urgency-type incontinence Analysis of covariance models were developed to examine change in incontinence frequency over 3 months. Results were summarized using least square mean estimates of changes in incontinence frequency in each group, as well as estimates of between-group difference in change in outcomes. Main efficacy analyses included all participants regardless of drop-out or adherence, consistent with an intention-to-treat principle. To address the potential for bias stemming from missing bladder diary data for up to 16% of participants who dropped out of interventions early, a multiple imputation procedure (SAS PROC MI, SAS Institute, Inc.) was used to impute values for data missing at follow-up. Imputation models included outcomes, randomization group, and baseline values.
Time Frame: Baseline and 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Episodes per day
Arm/Group | Yoga Therapy Group | Physical Conditioning Group
Number analyzed (Participants) | 28 | 28
Episodes per day | -1.7 [-2.6 to -0.91] | -1.7 [-2.6 to -0.7]
Statistical Analysis 1: Comparison: Yoga Therapy Group vs Physical Conditioning Group; Test type: Superiority; p = 0.89, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.2 to 1.3]

4. Secondary Outcome: Total Daytime Incontinence
Description: Change in frequency of total daytime incontinence Analysis of covariance models were developed to examine change in incontinence frequency over 3 months. Results were summarized using least square mean estimates of changes in incontinence frequency in each group, as well as estimates of between-group difference in change in outcomes. Main efficacy analyses included all participants regardless of drop-out or adherence, consistent with an intention-to-treat principle. To address the potential for bias stemming from missing bladder diary data for up to 16% of participants who dropped out of interventions early, a multiple imputation procedure (SAS PROC MI, SAS Institute, Inc.) was used to impute values for data missing at follow-up. Imputation models included outcomes, randomization group, and baseline values.
Time Frame: Baseline to 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Episodes per day
Arm/Group | Yoga Therapy Group | Physical Conditioning Group
Number analyzed (Participants) | 28 | 28
Episodes per day | -2.5 [-3.3 to -1.8] | -1.6 [-2.5 to -0.8]
Statistical Analysis 1: Comparison: Yoga Therapy Group vs Physical Conditioning Group; Test type: Superiority; p = 0.13, ANCOVA; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-0.3 to 2.0]

5. Secondary Outcome: Total Nighttime Incontinence
Description: Change in frequency of total nighttime incontinence Analysis of covariance models were developed to examine change in incontinence frequency over 3 months. Results were summarized using least square mean estimates of changes in incontinence frequency in each group, as well as estimates of between-group difference in change in outcomes. Main efficacy analyses included all participants regardless of drop-out or adherence, consistent with an intention-to-treat principle. To address the potential for bias stemming from missing bladder diary data for up to 16% of participants who dropped out of interventions early, a multiple imputation procedure (SAS PROC MI, SAS Institute, Inc.) was used to impute values for data missing at follow-up. Imputation models included outcomes, randomization group, and baseline values.
Time Frame: Baseline to 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Episodes per day
Arm/Group | Yoga Therapy Group | Physical Conditioning Group
Number analyzed (Participants) | 28 | 28
Episodes per day | -0.3 [-0.5 to -0.1] | -0.2 [-0.5 to 0.0]
Statistical Analysis 1: Comparison: Yoga Therapy Group vs Physical Conditioning Group; Test type: Superiority; p = 0.73, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.4]

6. Secondary Outcome: Incontinence Impact Questionnaire
Description: Change in questionnaire score for Incontinence Impact Questionnaire. Range 0-400, with higher scores mean worse function.
  Analysis of covariance models were developed to examine change in quality of life outcomes over 3 months. Results were summarized using least square mean estimates of changes in quality of life outcomes in each group, as well as estimates of between-group difference in change in outcomes. Main efficacy analyses included all participants regardless of drop-out or adherence, consistent with an intention-to-treat principle. To address the potential for bias stemming from missing bladder diary data for up to 16% of participants who dropped out of interventions early, a multiple imputation procedure (SAS PROC MI, SAS Institute, Inc.) was used to impute values for data missing at follow-up. Imputation models included outcomes, randomization group, and baseline values.
Time Frame: Baseline to 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Yoga Therapy Group | Physical Conditioning Group
Number analyzed (Participants) | 28 | 28
scores on scale | -74 [-103 to -45] | -94 [-127 to -60]
Statistical Analysis 1: Comparison: Yoga Therapy Group vs Physical Conditioning Group; Test type: Superiority; p = 0.38, ANCOVA; Mean Difference (Final Values) = -19.3, 95% CI 2-sided [-62.9 to 24.3]

7. Secondary Outcome: Urogenital Distress Inventory-6
Description: Change in the questionnaire score for Urogenital Distress Inventory-6. Range 0-100, with higher scores mean worse function.
  Analysis of covariance models were developed to examine change in quality of life outcomes over 3 months. Results were summarized using least square mean estimates of changes in quality of life outcomes in each group, as well as estimates of between-group difference in change in outcomes. Main efficacy analyses included all participants regardless of drop-out or adherence, consistent with an intention-to-treat principle. To address the potential for bias stemming from missing bladder diary data for up to 16% of participants who dropped out of interventions early, a multiple imputation procedure (SAS PROC MI, SAS Institute, Inc.) was used to impute values for data missing at follow-up. Imputation models included outcomes, randomization group, and baseline values.
Time Frame: Baseline to 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on scale
Arm/Group | Yoga Therapy Group | Physical Conditioning Group
Number analyzed (Participants) | 28 | 28
Scores on scale | -21 [-27 to -15] | -15 [-23 to -8]
Statistical Analysis 1: Comparison: Yoga Therapy Group vs Physical Conditioning Group; Test type: Superiority; p = 0.24, ANCOVA; Mean Difference (Final Values) = 5.6, 95% CI 2-sided [-3.7 to 14.8]

8. Secondary Outcome: Patient Perception of Bladder Condition
Description: Change in questionnaire score for Patient Perception of Bladder Condition. Range 1-6, with higher score mean worse function.
  Analysis of covariance models were developed to examine change in quality of life outcomes over 3 months. Results were summarized using least square mean estimates of changes in quality of life outcomes in each group, as well as estimates of between-group difference in change in outcomes. Main efficacy analyses included all participants regardless of drop-out or adherence, consistent with an intention-to-treat principle. To address the potential for bias stemming from missing bladder diary data for up to 16% of participants who dropped out of interventions early, a multiple imputation procedure (SAS PROC MI, SAS Institute, Inc.) was used to impute values for data missing at follow-up. Imputation models included outcomes, randomization group, and baseline values.
Time Frame: Baseline to 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Yoga Therapy Group | Physical Conditioning Group
Number analyzed (Participants) | 28 | 28
scores on scale | -1.3 [-1.7 to -0.8] | -1.0 [-1.5 to -0.5]
Statistical Analysis 1: Comparison: Yoga Therapy Group vs Physical Conditioning Group; Test type: Superiority; p = 0.46, ANCOVA; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.4 to 0.9]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Yoga Therapy Group | Physical Conditioning Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 17/28 | 14/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga Therapy Group (N=28) | Physical Conditioning Group (N=28)
Gastrointestinal Issues (Gastrointestinal disorders) | 0 (0) | 1 (1)
suspected prolapse (Renal and urinary disorders) | 1 (1) | 0 (0)
Broken Hand (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Eye soreness/sensitivity (Eye disorders) | 0 (0) | 1 (1)
Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upcoming Endoscopy For Small Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bursitis of left hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carpal Tunnel (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fall, Right arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot sprain at site of old fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
knee injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle or joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in right leg/foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right knee stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sciatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Severe right knee pain from previous injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thoracic pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Toe Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sprained ankle, hurt knee, and cracked patella (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
sprained wrist (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Mental Health Issues (Psychiatric disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Concussion (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Burst eardrum (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Macular Degeneration (Eye disorders) | 0 (0) | 1 (1)
Eye infection (Eye disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Cold (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Flu (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ear Infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT02342678/Prot_SAP_000.pdf